CLINICAL TRIAL: NCT03635944
Title: Nutritional Care Influences Head Growth at Discharge in Extremely Low Birth Weight Infants.
Brief Title: Nutritional Care and Head Growth in Preterm Infants
Acronym: KARLY
Status: Completed | Type: Observational
Sponsor: Hôpital de la Croix-Rousse (Other)
Responsible Party: Principal Investigator, Jean-charles PICAUD, MD, PhD, professor of pediatrics, Hôpital de la Croix-Rousse
Other Study IDs: PICAUD JC
Record Dates: First submitted 2018-08-14; First posted 2018-08-17 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Prematurity; Extreme; Growth Retardation
Keywords: growth; small for gestational age; prematurity; breastfeeding; fortification; parenteral nutrition; nutrition
MeSH Terms: conditions — Premature Birth; Breast Feeding; Hyperphagia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Infants born in Lyon (France)
- Group B: Infants born in Stockholm (Sweden)

SUMMARY:
As extremely low birth weight infants are high-risk patients, the study aimed to compare neonatal care, nutritional strategy and postnatal growth of these infants in two European neonatal units. A retrospective study included extremely low birth weight infants born in Lyon, France or in Stockholm, Sweden. Data on morbidity, treatments, care practices, macro-nutrient intakes and postnatal growth were collected to determine risk factors of extra uterine growth restriction at discharge.

By comparing postnatal growth in ELBW infants hospitalized in two European neonatal intensive care units with different nutritional and extra nutritional care,our objective was to evaluate the role of nutrition in this population of preterm infants.

DETAILED DESCRIPTION:
In a retrospective study, all ELBW infants (birth weight under 1000 g) with a gestational age between 23 and 28 weeks were included if they were admitted during the first 24 hours of life and stayed for at least seven weeks in two European units (Lyon, france, and Stockholm, Sweden). Parenteral and enteral nutrition policies were detailed and protein and energy intakes were collected.Growth assessment Postnatal growth was precisely evaluated and compared in the two groups of infants.

Body weight, crown-heel length and head circumference were measured in both units at birth and until discharge. We calculated z-scores and changes in z-scores between birth and 36 weeks post-conceptional age (delta z-score) for body weight, HC, and crown-to-heel length using Olsen's references. Intra-uterine growth restriction was defined as a birth weight below or equal to minus two standard deviations. Extra-uterine growth restriction was defined as a z-score loss above or equal one standard deviation between birth and 36 weeks PCA. I

ELIGIBILITY:
Inclusion Criteria:

* birth weight under 1000 grams
* gestational age (GA) between 23 and 28 weeks
* born in 2012
* admitted during the first 24 hours of life
* stayed in one of the two studied units for at least 7 weeks before transfer to the referring hospital, discharge to home or death.

Exclusion Criteria:

* Neonates with congenital anomalies

Ages: 1 Minute to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Extremely low birth weight infants born in two European tertiary care centres: neonatal unit of Croix Rousse Hospital in Lyon, France and the neonatal unit of Astrid Lindgren Children's Hospital in Stockholm, Sweden
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Weight gain during hospitalization | between birth and 40 weeks
  difference in weight between birth and discharge

SECONDARY OUTCOMES:
Crown-heel length gain during hospitalization | between birth and 40 weeks
  difference in recumbent length between birth and discharge
Head circumference gain during hospitalization | between birth and 40 weeks
  difference in head circumference between birth and discharge

CONTACTS AND LOCATIONS:
Overall Officials: jean-charles picaud, MD, PhD, Principal Investigator — Hopital de la croix rousse
Locations (1):
- Hopital de la croix rousse, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided